CLINICAL TRIAL: NCT04711603
Title: A Phase III Clinical Study of MR13A9 in Hemodialysis Patients With Pruritus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MR13A9-5
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2023-04

CONDITIONS: Uremic Pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MR13A9/MR13A9 (Experimental): Patients are administered MR13A9 for 6 weeks (double-blind period), followed by MR13A9 for 52 weeks (open-label period).
  Interventions: Drug: MR13A9
- Placebo/MR13A9 (Placebo Comparator): Patients are administered Placebo for 6 weeks (double-blind period), followed by MR13A9 for 52 weeks (open-label period).
  Interventions: Drug: MR13A9; Drug: Placebo

INTERVENTIONS:
Drug: MR13A9 — Intravenous administration
Drug: Placebo — Intravenous administration
  Arms: Placebo/MR13A9

SUMMARY:
Double-blind, Placebo-controlled study to confirm the superiority of MR13A9 to placebo, and followed by extension, open-label treatment to confirm long-term safety of MA13A9 in hemodialysis patients with pruritus.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Chronic Kidney Disease (CKD) has been on hemodialysis 3 times per week
* Patient receiving treatment for itch
* Patient has a baseline NRS score > 4

Exclusion Criteria:

* Patient has pruritus cause other than CKD or its complications
* Patients has hepatic cirrhosis
* Patient has a known history of allergic reaction to opiates

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2021-01-16 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshitaka Shimizu, Study Director — Kissei Pharmaceutical Co., Ltd.
Locations (1):
- Research Site, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Narita I, Tsubakihara Y, Takahashi N, Ebata T, Uchiyama T, Marumo M, Okamura S, Gejyo F; MR13A9-5 Trial Investigators. Difelikefalin for Hemodialysis Patients with Pruritus in Japan. NEJM Evid. 2023 Nov;2(11):EVIDoa2300094. doi: 10.1056/EVIDoa2300094. Epub 2023 Oct 17. PMID 38320524

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two hundred thirty subjects were screened. A total of 178 subjects included in the study and were randomly assigned to the study drug. The number of subjects in the double-blind period (6 weeks) was 178. The number of subjects who transitioned to the extension period (52 weeks) was 168. The number of subjects who completed Week 58 was 122.
Pre-assignment Details: Previously treated hemodialysis patients with pruritus were enrolled in a 1:1 ratio to either MR13A9 0.5 μg/kg group or Placebo group. Subjects who received placebo in the double-blind period received MR13A9 0.5 μg/kg in the extension period.
Groups:
- Double Blind Period: MR13A9 0.5 μg/kg Group: MR13A9 was injected into the venous line of the dialysis circuit at the end of each dialysis session for 6 weeks (3 times weekly, 18 times in total).
  The dose of the study drug was determined according to mentioned below based on the subject's dry weight before dialysis on the start day of the screening period.
  1. <45.0 kg: 17.5 μg
  2. >=45.0 kg, <65.0 kg: 25.0 μg
  3. >=65.0 kg, <85.0 kg: 35.0 μg
  4. >=85.0 kg: 42.5 μg
- Double Blind Period: Placebo Group: Placebo was injected into the venous line of the dialysis circuit at the end of each dialysis session for 6 weeks (3 times weekly, 18 times in total).
  The dose of the study drug was determined according to mentioned below based on the subject's dry weight before dialysis on the start day of the screening period.
  1. <45.0 kg: 0 μg
  2. >=45.0 kg, <65.0 kg: 0 μg
  3. >=65.0 kg, <85.0 kg: 0 μg
  4. >=85.0 kg: 0 μg
- Entire Study: MR13A9/MR13A9 Group: [Double-blind period (6 weeks)] The subjects in this group received the investigational drug for 6 weeks as the MR13A9 0.5 μg/kg group.
  [Extension period (52 weeks)] The study drug was injected into the venous line of the dialysis circuit at the end of each dialysis session for 52 weeks (3 times weekly, 156 times in total).
  The dose of the study drug was determined according to mentioned below, and the dose of the study drug from Week 6 to immediately before Week 34 will be determined based on the subject's dry weight before dialysis at Week 6. The dose of the study drug after Week 34 will be determined based on the subject's dry weight before dialysis at Week 34. The study drug (MR13A9) will not be administered at Week 58.
  1. <45.0 kg: 17.5 μg
  2. >=45.0 kg, <65.0 kg: 25.0 μg
  3. >=65.0 kg, <85.0 kg: 35.0 μg
  4. >=85.0 kg: 42.5 μg
- Entire Study: Placebo/MR13A9 Group: [Double-blind period (6 weeks)] The subjects in this group received the investigational drug for 6 weeks as the Placebo group.
  [Extension period (52 weeks)] The study drug was injected into the venous line of the dialysis circuit at the end of each dialysis session for 52 weeks (3 times weekly, 156 times in total).
  The dose of the study drug was determined according to mentioned below, and the dose of the study drug from Week 6 to immediately before Week 34 will be determined based on the subject's dry weight before dialysis at Week 6. The dose of the study drug after Week 34 will be determined based on the subject's dry weight before dialysis at Week 34. The study drug (MR13A9) will not be administered at Week 58.
  1. <45.0 kg: 17.5 μg
  2. >=45.0 kg, <65.0 kg: 25.0 μg
  3. >=65.0 kg, <85.0 kg: 35.0 μg
  4. >=85.0 kg: 42.5 μg
Period: Double-blind Period (6 Weeks)
Arm/Group | Double Blind Period: MR13A9 0.5 μg/kg Group | Double Blind Period: Placebo Group | Entire Study: MR13A9/MR13A9 Group | Entire Study: Placebo/MR13A9 Group
Started | 89 | 89 | 0 | 0
Completed | 85 | 83 | 0 | 0
Not Completed | 4 | 6 | 0 | 0
Not completed — Adverse Event | 4 | 3 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — 4 consecutive missed doses of the study drug | 0 | 1 | 0 | 0
Period: Extension Period (52 Weeks)
Arm/Group | Double Blind Period: MR13A9 0.5 μg/kg Group | Double Blind Period: Placebo Group | Entire Study: MR13A9/MR13A9 Group | Entire Study: Placebo/MR13A9 Group
Started | 0 | 0 | 85 | 83
Completed | 0 | 0 | 68 | 54
Not Completed | 0 | 0 | 17 | 29
Not completed — Adverse Event | 0 | 0 | 6 | 18
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 5
Not completed — 7 consecutive missed doses of the study drug | 0 | 0 | 5 | 2
Not completed — Needed to prioritize the treatment of adverse events | 0 | 0 | 0 | 1
Not completed — Difficulty in using iPad for efficacy evaluation | 0 | 0 | 0 | 1
Not completed — The input rate of the symptom diary was low and no improvement | 0 | 0 | 0 | 1
Not completed — Transferred to another hospital | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- MR13A9 0.5 μg/kg Group: The study drug was injected into the venous line of the dialysis circuit at the end of each dialysis session for 6 weeks (3 times weekly, 18 times in total).
  The dose of the study drug (MR13A9) was determined according to mentioned below based on the subject's dry weight before dialysis on the start day of the screening period.
  1. <45.0 kg: 17.5 μg
  2. >=45.0 kg, <65.0 kg: 25.0 μg
  3. >=65.0 kg, <85.0 kg: 35.0 μg
  4. >=85.0 kg: 42.5 μg
- Placebo Group: The study drug was injected into the venous line of the dialysis circuit at the end of each dialysis session for 6 weeks (3 times weekly, 18 times in total).
- Total: Total of all reporting groups
Arm/Group | MR13A9 0.5 μg/kg Group | Placebo Group | Total
Number analyzed (Participants) | 85 | 88 | 173
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 36 | 76
  >=65 years | 45 | 52 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (10.5) | 64.1 (12.7) | 64.2 (11.7)
Age, Customized [Median (Inter-Quartile Range); unit: years] | 66 [57 to 72] | 67 [58 to 73] | 66 [57 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 27
  Male | 74 | 72 | 146
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 85 | 88 | 173
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 85 | 88 | 173
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 85 | 88 | 173
Dry Weight at the start of Screening [Mean (Standard Deviation); unit: kg] | 62.64 (11.63) | 63.33 (12.94) | 62.99 (12.28)
Hemodialysis History [Mean (Standard Deviation); unit: years] | 8.4 (7.6) | 7.9 (6.7) | 8.1 (7.1)
Disease Duration of Itch [Mean (Standard Deviation); unit: years] | 5.7 (5.5) | 4.6 (3.8) | 5.1 (4.7)
Average NRS Score [Mean (Standard Deviation); unit: points] — Looking back on the period between the time of awakening on the previous day of assessment and the time of awakening on the day of assessment (including sleeping hours) once daily, subjects will assess the NRS score for the most severe itching by themselves. The most severe itching within the day will be assessed in integer on a scale ranging from 0 to 10, where 0 represents no itching and 10 represents worst itching imaginable.
  points | 6.57 (1.29) | 6.40 (1.28) | 6.48 (1.28)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Mean NRS Score at Week 4
Description: The change from baseline in the mean NRS score at each time point was calculated using an MMRM with the change from baseline in the mean NRS score at each time point as an objective variable, group, time point, and group-by-time point interaction as fixed effects, mean NRS score at baseline and presence or absence of prior treatment with nalfurafine hydrochloride as dynamic allocation factors as a covariate, and subjects as a random effect for data up to Week 4 of the double-blind period in FAS.
  Looking back on the period between the time of awakening on the previous day of assessment and the time of awakening on the day of assessment (including sleeping hours) once daily, subjects will assess the NRS score for the most severe itching by themselves. The most severe itching within the day will be assessed in integer on a scale ranging from 0 to 10, where 0 represents no itching and 10 represents worst itching imaginable.
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: points
Arm/Group | MR13A9 0.5 μg/kg Group | Placebo Group
Number analyzed (Participants) | 85 | 88
points | -2.06 (0.20) | -1.09 (0.20)
Statistical Analysis 1: Comparison: MR13A9 0.5 μg/kg Group vs Placebo Group; Test type: Superiority; p < 0.001, MMRM; Placebo difference = -0.97, 95% CI 2-sided [-1.52 to -0.42], Standard Error of Mean 0.28

ADVERSE EVENTS:
Time Frame: Up to Week 58 (6-week Double Blind Treatment Period and 52-week Extension Period)
Description: Adverse Events were not collected separately for the Extension Period, but rather were pre-specified to be collected for the separate "MR-MR Group" and "P-MR Group" Arms/Groups separately for the Double Blind Period and for the entire study. Therefore, we have presented separate Arms/Groups for the Double-Blind Period (data monitored/assessed over 6 weeks), and the Entire Study Period (data monitored/assessed over 58 weeks)
Groups:
- Entire Study: MR-MR Group: [Double-blind period (6 weeks)] The subjects in this group received the investigational drug for 6 weeks as the MR13A9 0.5 μg/kg group.
  [Extension period (52 weeks)]
  The study drug was injected into the venous line of the dialysis circuit at the end of each dialysis session for 52 weeks (3 times weekly, 156 times in total).
  The dose of the study drug was determined according to mentioned below, and the dose of the study drug from Week 6 to immediately before Week 34 will be determined based on the subject's dry weight before dialysis at Week 6. The dose of the study drug after Week 34 will be determined based on the subject's dry weight before dialysis at Week 34. The study drug (MR13A9) will not be administered at Week 58.
  1. <45.0 kg: 17.5 μg
  2. >=45.0 kg, <65.0 kg: 25.0 μg
  3. >=65.0 kg, <85.0 kg: 35.0 μg
  4. >=85.0 kg: 42.5 μg
- Entire Study: P-MR Group: [Double-blind period (6 weeks)] The subjects in this group received the investigational drug for 6 weeks as the Placebo group.
  [Extension period (52 weeks)]
  The study drug was injected into the venous line of the dialysis circuit at the end of each dialysis session for 52 weeks (3 times weekly, 156 times in total).
  The dose of the study drug was determined according to mentioned below, and the dose of the study drug from Week 6 to immediately before Week 34 will be determined based on the subject's dry weight before dialysis at Week 6. The dose of the study drug after Week 34 will be determined based on the subject's dry weight before dialysis at Week 34. The study drug (MR13A9) will not be administered at Week 58.
  1. <45.0 kg: 17.5 μg
  2. >=45.0 kg, <65.0 kg: 25.0 μg
  3. >=65.0 kg, <85.0 kg: 35.0 μg
  4. >=85.0 kg: 42.5 μg
Arm/Group | Double Blind Period: MR13A9 0.5 μg/kg Group | Double Blind Period: Placebo Group | Entire Study: MR-MR Group | Entire Study: P-MR Group
All-Cause Mortality (participants affected / at risk) | 0/89 | 1/89 | 2/85 | 2/83
Serious Adverse Events (participants affected / at risk) | 7/89 | 10/89 | 33/85 | 38/83
Other Adverse Events (participants affected / at risk) | 27/89 | 24/89 | 74/85 | 74/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Blind Period: MR13A9 0.5 μg/kg Group (N=89) | Double Blind Period: Placebo Group (N=89) | Entire Study: MR-MR Group (N=85) | Entire Study: P-MR Group (N=83)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paroxysmal atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Renal cyst infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shunt infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract operation complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shunt aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Shunt occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 6 (6) | 4 (6)
Shunt stenosis (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 2 (7) | 7 (18)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Large intestinal polypectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (4)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Blind Period: MR13A9 0.5 μg/kg Group (N=89) | Double Blind Period: Placebo Group (N=89) | Entire Study: MR-MR Group (N=85) | Entire Study: P-MR Group (N=83)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1) | 12 (13) | 8 (11)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (4) | 11 (18) | 18 (26)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 7 (16) | 5 (6)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 8 (8) | 3 (5)
Pyrexia (General disorders) | 4 (4) | 3 (3) | 15 (17) | 18 (20)
Vaccination site pain (General disorders) | 1 (1) | 0 (0) | 5 (6) | 5 (7)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 5 (5) | 3 (3)
Nasopharyngitis (Infections and infestations) | 3 (4) | 2 (2) | 13 (25) | 15 (22)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 15 (20) | 7 (8)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 5 (8) | 6 (8)
Shunt stenosis (Injury, poisoning and procedural complications) | 5 (5) | 0 (0) | 11 (15) | 8 (16)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 8 (12) | 12 (18)
Vaccination complication (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 14 (19) | 12 (17)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3) | 5 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 8 (9) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 11 (11) | 10 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 4 (5) | 9 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 9 (10) | 8 (12)
Dizziness (Nervous system disorders) | 0 (0) | 3 (4) | 5 (7) | 9 (11)
Headache (Nervous system disorders) | 2 (3) | 0 (0) | 6 (8) | 10 (14)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 5 (6) | 6 (6)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 6 (6) | 7 (10)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 5 (7) | 3 (5)
Dialysis hypotension (Vascular disorders) | 0 (0) | 1 (1) | 3 (9) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT04711603/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT04711603/SAP_001.pdf